CLINICAL TRIAL: NCT04799990
Title: Post-Marketing Real World Safety Study of Risankizumab in the United States
Brief Title: Study to Assess Adverse Events When Subcutaneous Risankizumab Injection is Given to Adult Participants With Psoriasis in Real World Setting
Status: Withdrawn | Type: Observational
Why Stopped: Study is not recruiting and using secondary data sources only
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P16-772
Record Dates: First submitted 2021-03-15; First posted 2021-03-16 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — risankizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Risankizumab: Participants will receive risankizumab as prescribed by their physician.
  Interventions: Drug: Risankizumab
- Comparator Group 1: Participants will receive biologics other than interleukin (IL)-23 antagonists as prescribed by their physician.
  Interventions: Biological: Comparator 1
- Comparator Group 2: Participants will receive non-biologic systemic small molecules as prescribed by their physician.
  Interventions: Drug: Comparator 2

INTERVENTIONS:
Drug: Risankizumab — Subcutaneous Injection
  Other Names: Skyrizi
  Groups: Risankizumab
Biological: Comparator 1 — Subcutaneous or Intravenous Injection
  Groups: Comparator Group 1
Drug: Comparator 2 — Oral, Opthalmic, Subcutaneous or Intravenous Injection
  Groups: Comparator Group 2

SUMMARY:
Study is not recruiting and using secondary data sources only

DETAILED DESCRIPTION:
Study is not recruiting and using secondary data sources only

ELIGIBILITY:
Study is not recruiting and using secondary data sources only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study is not recruiting and using secondary data sources only
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Incidence Rate of Participants With Major Adverse Cardiovascular Events (MACE) | Up to approximately 10 years
  MACE is defined as any fatal or nonfatal myocardial infarction (MI) or stroke (including cerebral infarction, nontraumatic intracerebral hemorrhage, and nontraumatic subarachnoid hemorrhage).

SECONDARY OUTCOMES:
Incidence Rate of Participants With Serious Infections | Up to approximately 10 years
  Serious infections is defined as inpatient encounter for infections or receiving treatment with intravenous antibiotics, anti-viral or anti-fungal medications.
Incidence Rate of Participants With Tuberculosis | Up to approximately 10 years
  Tuberculosis is defined as inpatient encounter for active tuberculosis, or outpatient encounter with a dispensing of at least two classes of first-line anti-tuberculosis medications (e.g., isoniazid, rifampin, pyrazinamide, or ethambutol) for a sufficient duration to differentiate prophylaxis and treatment use.
Incidence Rate of Participants With Opportunistic Infections Excluding Tuberculosis and Herpes Zoster | Up to approximately 10 years
  Opportunistic infections are defined as outpatient or inpatient encounter for opportunistic infections excluding tuberculosis and herpes zoster.
Incidence Rate of Participants With Serious Hypersensitivity Reactions | Up to approximately 10 years
  Serious hypersensitivity reactions are defined as emergency department (ED) or inpatient encounter for serious hypersensitivity reactions including anaphylaxis.
Incidence Rate of Participants With Autoimmune Disease | Up to approximately 10 years
  Autoimmune disease is defined as outpatient or inpatient encounter for systemic lupus erythematosus (SLE).
Incidence Rate of Participants With Neurologic or Demyelinating Disease | Up to approximately 10 years
  Neurologic or demyelinating disease is defined as outpatient or inpatient encounter for multiple sclerosis (MS), optic neuritis, and the peripheral demyelinating disease Guillain-Barré syndrome.
Incidence Rate of Participants With Gastrointestinal Adverse Events | Up to approximately 10 years
  Gastrointestinal adverse events are defined as inpatient encounter for gastrointestinal perforation. Gastrointestinal (GI) perforation is defined as perforation of the esophagus, stomach, small intestine, large intestine, and unspecified lower GI.
Incidence Rate of Participants With Nonmalignant-Hematologic Adverse Events | Up to approximately 10 years
  Nonmalignant-hematologic adverse events are defined as outpatient or inpatient encounter for a non-malignant hematological adverse events (pancytopenia, agranulocytosis and aplastic anemia).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided